CLINICAL TRIAL: NCT04894474
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Parallel-group, Group-sequential Study to Evaluate Efficacy, Safety and Tolerability of BI 767551 for Post-exposure Prevention of SARS-CoV-2 Infection in Household Contacts to a Confirmed SARS-CoV-2 Infected Individual
Brief Title: A Study to Test Whether BI 767551 Can Prevent COVID-19 in People Who Have Been Exposed to SARS-CoV-2
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: project terminated
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1487-0003; 2021-000408-39 (EudraCT Number)
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 767551 inhalation and placebo intravenous infusion (Experimental)
  Interventions: Drug: BI 767551 inhalation; Drug: Placebo intravenous
- BI 767551 intravenous infusion and placebo inhalation (Experimental)
  Interventions: Drug: BI 767551 intravenous; Drug: Placebo inhalation
- Placebo inhalation and placebo intravenous infusion (Placebo Comparator)
  Interventions: Drug: Placebo intravenous; Drug: Placebo inhalation

INTERVENTIONS:
Drug: BI 767551 intravenous — BI 767551 intravenous
  Arms: BI 767551 intravenous infusion and placebo inhalation
Drug: BI 767551 inhalation — BI 767551 inhalation
  Arms: BI 767551 inhalation and placebo intravenous infusion
Drug: Placebo intravenous — Placebo intravenous
  Arms: BI 767551 inhalation and placebo intravenous infusion; Placebo inhalation and placebo intravenous infusion
Drug: Placebo inhalation — Placebo inhalation
  Arms: BI 767551 intravenous infusion and placebo inhalation; Placebo inhalation and placebo intravenous infusion

SUMMARY:
This study is open to adults living with a person who has tested positive for the coronavirus SARS-CoV-2. People who do not have symptoms of COVID-19 can take part in this study. The study is done to find out whether a medicine called BI 767551 can prevent COVID-19. BI 767551 is an antibody against the coronavirus SARS-CoV-2.

Participants are put into 3 groups randomly, which means by chance.

* 1 group gets BI 767551 via an inhaler and placebo as an infusion
* 1 group gets BI 767551 as an infusion and placebo via an inhaler
* 1 group gets placebo both via an inhaler and as an infusion

All participants get study medicine once at study start and after 1 week. Placebo inhaler and infusion look like BI 767551 inhaler and infusion but do not contain any medicine.

Participants are in the study for about 3 months. During this time, they visit the study site about 10 times. About 7 of the 10 visits can be done at the participant's home. Participants are regularly tested for the coronavirus SARS-CoV-2. The doctors check whether the participants have been infected with the coronavirus and whether they have symptoms. The results are compared between the treatment groups. The doctors check the health of the participants and note any health problems that could have been caused by BI 767551.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, males and females
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Asymptomatic for Coronavirus Disease 2019 (COVID-19) at time of screening and at randomization
* Household contact with exposure to an individual with a diagnosis of Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (i.e. exposure to the index case)
* Randomization within 96 hours of collection of the index cases' positive SARS-CoV-2 diagnostic test sample (nucleic acid or antigen-based) from any respiratory tract specimen (e.g. oropharyngeal, nasopharyngeal (NP), or nasal swab, or saliva); based on test sample collection date, not the result date.
* From screening and randomization, the trial participant anticipates living in the same household with the index case until protocol Day 29.
* Women of childbearing potential (WOCBP)* and men able to father a child must be ready and able to use highly effective methods of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

  * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 24 months without an alternative medical cause.

Exclusion Criteria:

* Body weight of less than 40 kg
* Residents of skilled nursing facilities. Definition of skilled nursing facility: assisted living facility that typically provides daily nursing care, 24-hour supervision, three meals a day, and assistance with everyday activities.
* History of laboratory confirmed SARS-CoV-2 infection (e.g. antigen or nucleic acid test)at any time before screening
* Active respiratory or non-respiratory symptoms consistent with COVID-19, in the opinion of the investigator
* History of respiratory or non-respiratory symptoms consistent with COVID-19, within the prior 6 months to screening, in the opinion of the investigator
* Participant has lived with individuals who have had previous SARS-CoV-2 infection or currently lives with individuals who have SARS-CoV-2 infection, with the exception of the index case(s) who is defined as the first individual(s) known to be infected in the household
* Receipt of intravenous immunoglobulin within 12 weeks prior to Visit 2
* Receipt of COVID-19 convalescent plasma treatment at any time prior to Visit 2
* Receipt of any SARS-CoV-2 monoclonal antibody treatment at any time prior to Visit 2
* Receipt of SARS-CoV-2 vaccine at any time prior to Visit 2
* Receipt of an investigational product for COVID-19 within 5 half-lives prior to Visit 2
* Receipt of systemic steroids (e.g. prednisone, dexamethasone) within 4 weeks prior to Visit 2 unless used for chronic condition
* Subjects who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Any co-morbidity requiring surgery within 7 days prior to study entry, or that is considered life threatening in the opinion of investigator within 30 days prior to randomization
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study
* Subjects not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the subject an unreliable trial participant)
* Currently enrolled in any other type of medical research judged not to be compatible with this study
* Known allergy/sensitivity or any hypersensitivity to any of the components used in the formulation of the interventions
* Previous enrolment in this trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-17 (Estimated); Primary Completion 2022-05-23 (Estimated); Study Completion 2022-07-24 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is symptomatic SARS-CoV-2 infection (RT-qPCR confirmed based on NP swabs, with a score >= 2 on the WHO Clinical Progression Scale) (Cohort A only) | up to 31 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
  qPCR: Quantitative Reverse Transcription Polymerase chain reaction; WHO: World Health Organisation;
  The 11-point WHO Clinical Progression Scale ranges from 0 to 10, with a higher score indicating a worsening of the symptoms.

SECONDARY OUTCOMES:
SARS-CoV-2 infection, with or without symptoms (Cohort A only) | up to 31 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Asymptomatic SARS-CoV-2 infection (with a score not exceeding 1 on the WHO Clinical Progression Scale) (Cohort A only) | up to 31 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Severity of COVID-19 (No, mild, moderate, or severe COVID-19, with a maximum score of 0, 1-3, 4-5, or >= 6,respectively, on the WHO Clinical Progression Scale) (Cohort A) | up to 98 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Severity of COVID-19 (No, mild, moderate, or severe COVID-19, with a maximum score of 0, 1-3, 4-5, or >= 6,respectively, on the WHO Clinical Progression Scale) (Cohort B) | up to 98 days
  Cohort B: positive SARS-CoV-2 RT-qPCR test* or positive serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Hospitalization due to COVID-19 for >= 24 hours (Cohort A) | up to 98 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Hospitalization due to COVID-19 for >= 24 hours (Cohort B) | up to 98 days
  Cohort B: positive SARS-CoV-2 RT-qPCR test* or positive serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Hospitalization due to COVID-19 for >= 24 hours or death (Cohort A) | up to 98 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Hospitalization due to COVID-19 for >= 24 hours or death (Cohort B) | up to 98 days
  Cohort B: positive SARS-CoV-2 RT-qPCR test* or positive serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Death (Cohort A) | up to 98 days
  Cohort A: negative SARS-CoV-2 RT-qPCR* and serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.
Death (Cohort B) | up to 98 days
  Cohort B: positive SARS-CoV-2 RT-qPCR test* or positive serology test* at baseline.
  *test result from day of dosing (baseline) will be retrospectively determined by the sponsor-provided central laboratory. The designation of Cohorts is used only for the analysis not randomization.

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: Related Info — http://www.mystudywindow.com/